CLINICAL TRIAL: NCT05128682
Title: The Effect Of Acute Pudendal Nerve Stimulation On Leak Point Pressure In Women Urodynamic: Early Feasibility Study
Brief Title: Acute Pudendal Nerve Stimulation On Leak Point Pressure In Women Urodynamic Early Feasibility Study
Acronym: PNS_UDT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This is an early feasibility study. After the first 4 patients completed study activities, the investigator determined that this protocol is not the best way to test the study hypothesis.
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-286
Record Dates: First submitted 2021-09-22; First posted 2021-11-22 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Urinary Incontinence
Keywords: pudendal nerve; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Subjects who meet all eligibility criteria will be enrolled in the study and will undergo urodynamic testing with UPP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Urodynamic testing with and without pudendal nerve stimulation (Other): The neuromodulation settings of the implanted device will be adjusted to deliver acute simulation. Urodynamic testing (UDT) will be completed by filling the bladder and observing for urinary leakage. The assessment will be completed with the stimulation sets turned off and then turned on. At the end of the UDT the settings will be returned to the previously set therapeutic values. The neuromodulation settings constitute the "dose" and can include the voltage/current amplitude, frequency, pulse width, on time/off time duration and electrode polarity assignments. These parameters are limited by the available ranges of the approved neurostimulation device and will be adjusted during the study by the principal investigator to stay within the safe and comfortable levels for each individual study subject.
  Interventions: Diagnostic Test: Urodynamic testing with and without pudendal nerve stimulation

INTERVENTIONS:
Diagnostic Test: Urodynamic testing with and without pudendal nerve stimulation — A urodynamic test (UDT) for eligible subjects with and without acute PNS will be conducted. Prior to introducing the acute PNS, the subject's original stimulation properties will be turned off. The implanted neurostimulator device will be programmed to deliver acute PNS per individual tolerance level with the objective of increasing external urethral sphincter pressure. The LPP during Valsalva maneuver or forceful coughing will be assessed with and without acute PNS. The LPP will be assessed at increasing bladder volumes until major detrusor instability, significant leakage (more than drops, stream) or subject discomfort (strong desire to void) is observed. Finally, a UPP with PNS set in an on/off cycling regimen will be conducted to observe the effect on pressures along the length of the urethra.

SUMMARY:
The purpose of this study is tp evaluate the changes in stress induced Urethral Leak Point Pressures (LPP) and other urodynamic measurements in response to acute pudendal nerve stimulation (PNS) in patients with a pre-existing implanted urological neurostimulator stimulating the pudendal nerve.

DETAILED DESCRIPTION:
Patients with a neurostimulator implanted at the pudendal nerve will be enrolled and undergo urodynamic testing. Before testing, study staff will provide an oral antibiotic (to reduce the risk of infection) and adjust the stimulation settings with a goal to increase urethral pressure from baseline by at lest 20cm H2O, without causing the patient discomfort/distress. These settings will be used throughout urodynamics. Before filling the bladder, a urethral pressure profile study will be completed 3 times with stimulation off, then 3 times with stimulation on. Leak point pressure (LPP) testing will then be completed. The patient's bladder will be filled following standard urodynamic testing protocol. Filling will be paused every 50-100mL to complete LPP assessment. Subjects will be asked to complete a light cough, medium cough, forceful cough, and Valsalva maneuver (in that order). Detrusor pressure will be measured at each event, and staff will document whether or not a leak was elicited. This will be completed with stimulation off, then with stimulation on, as the bladder is filled. Once the subject reports a strong urge to void, urethral pressure profile assessment will be completed again: 3 times with stimulation off, then 3 times with stimulation on. Once urodynamic testing is complete and the patient's bladder is emptied, a measurement of urethral pressure will be completed with stimulation off, then during 5 seconds of stimulation, then again with stimulation off.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 85 years old, inclusive.
* Implanted with a neurostimulation device for at least 3 months prior to consent (Medtronic Interstim neurostimulator models 3023, 3058, 97810, or similar).
* Implanted with a tined lead that is placed and functionable at the pudendal nerve (Medtronic model 3889 or similar).
* Is capable of understanding clinical study procedures and giving informed consent.
* Willing and able to visit the clinic for the UDT evaluation (study procedure)

Exclusion Criteria:

* Medically unstable at time of study and unsafe to undergo urodynamic testing as determined by the investigator.
* History of bladder cancer.
* History of pelvic radiotherapy.
* Active gross hematuria.
* Active symptomatic urinary tract infection (UTI)
* Active symptomatic uncontrolled bladder instability as determined by the investigator.
* History or symptoms of cystocele, enterocele, or rectocele of grade 3 or 4. Per the medical record or as determined by the investigator.
* Presence of an artificial urinary sphincter.
* Women who are pregnant and/or have given birth in the previous 12 months
* Any medical condition that would interfere with the patient's ability to comply with the protocol and/or may affect the outcome of this study or safety of the subject as determined by the investigator
* BMI greater than 39.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Beaumont Hospital - Royal Oak
Locations (2):
- United States (2):
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Beaumont Hospital Royal Oak, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Urodynamic Testing With and Without Pudendal Nerve Stimulation: A urodynamic test (UDT) for eligible subjects with and without acute PNS will be conducted. Prior to introducing the acute PNS, the subject's original stimulation properties will be turned off. The implanted neurostimulator device will be programmed to deliver acute PNS per individual tolerance level with the objective of increasing external urethral sphincter pressure. UDT will be completed by filling the bladder and observing for urinary leakage. The LPP during Valsalva maneuver or forceful coughing will be assessed with and without acute PNS. The LPP will be assessed at increasing bladder volumes until major detrusor instability, significant leakage (more than drops, stream) or subject discomfort (strong desire to void) is observed. Finally, a UPP with PNS set in an on/off cycling regimen will be conducted to observe the effect on pressures along the length of the urethra.
Period: Overall Study
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Females with a neurostimulator implanted device
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [41 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Pulse Amplitude Triggering Patient Sensation at First Verbally Reported Sensation.
Description: PNS final settings including: pulse amplitude, measured in mA, when subject first verbalizes sensation. Pulse amplitude is the amplitude of the electric pulses; measured in Milliamps (mA). This is a setting present on the neuromodulation device, it is not calculated.
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Population: One subject did not have a pulse amplitude recorded.
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 3
mA | 0.76 (0.45)

2. Primary Outcome: Pulse Frequency Triggering Patient Sensation at First Verbally Reported Sensation.
Description: PNS final settings including: pulse frequencies, measured in Hz, when subject first verbalizes sensation.
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 4
Hz | 45 (20.18)

3. Primary Outcome: Pulse Width Triggering Patient Sensation at First Verbally Reported Sensation.
Description: PNS final settings including: pulse widths, measured in µs, when the subject first verbalizes sensation.
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Population: One participant did not have a pulse width recorded
Measure: Mean (Standard Deviation); unit: µs
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 3
µs | 210 (0)

4. Primary Outcome: Identification of All Study-related Adverse Events
Description: Safety and tolerability will be assessed in relation to the incidence of study related adverse events reported.
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 4
Participants | 0

5. Primary Outcome: Changes in Leak Point Pressure (LPP) Upon Acute PNS
Description: Measurement of the change in LPP with acute PNS compared to without stimulation. To assess LPP, the urethral pressure increase will be calculated by subtracted pressure with and without stimulation at the "final setting". In cm water.
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Population: No leaks were noted in any of the four participants.
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 0

6. Secondary Outcome: Effect of Acute PNS on the Urethral Pressure Profile (UPP).
Description: Measure the maximum urethral closure pressure with and without programmed pudendal nerve stimulation. In cm water.
  Urethral pressure profile is a test of the bladder neck, urethra, and urethral sphincters that is completed with urodynamic equipment. A small catheter is pulled at a constant rate from the bladder neck down the urethra to provide the functional length of the urethra and points of maximal urethral resistance at the urethral sphincter. It is a procedure used to measure the competency of the urethral sphincter (outflow resistance).
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Population: Two participants did not complete.
Measure: Mean (Standard Deviation); unit: cm water
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 2
cm water
  Max Urethral Closure Pressure With Stimulation | 53.9 (4.21)
  Max Urethral Closure Pressure No Stimulation | 51.2 (3.08)

7. Secondary Outcome: Effect of Acute PNS on Max Cystometic Capacity.
Description: Max cystometic capacity will be collected, with and without programmed PNS, the difference will be reported. In mL.
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Population: Not collected on any participants due to testing limitations.
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 0

8. Secondary Outcome: Effect of Acute PNS on Post Void Residual.
Description: Post void residual collected at end of UDT testing. Measured in mL.
Time Frame: After Visit 2 activities are complete. An average of 30 days after enrollment.
Population: Three participants did not have data collected.
Measure: Number; unit: mL
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
Number analyzed (Participants) | 1
mL | 30

ADVERSE EVENTS:
Time Frame: This was collected over approximately 5 weeks, from initial consent to subject study completion.
Groups:
- Urodynamic Testing With and Without Pudendal Nerve Stimulation: The neuromodulation settings of the implanted device will be adjusted to deliver acute simulation. Urodynamic testing (UDT) will be completed by filling the bladder and observing for urinary leakage. The assessment will be completed with stimulation turned off and on. At the end of the UDT the settings will be returned to the previously settings.
  Urodynamic testing with and without pudendal nerve stimulation: A urodynamic test (UDT) with and without acute PNS will be conducted. Prior to introducing the acute PNS, the subject's original stimulation properties will be turned off. The implanted neurostimulator device will be programmed to deliver acute PNS per individual tolerance level with the objective of increasing external urethral sphincter pressure. The LPP will be assessed with and without acute PNS. The LPP will be assessed at increasing bladder volumes until major detrusor instability, significant leakage (more than drops, stream) or subject discomfort (strong desire to void) is observed. Finally, a UPP with PNS set in an on/off cycling regimen will be conducted to observe the effect on pressures along the length of the urethra.
Arm/Group | Urodynamic Testing With and Without Pudendal Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
After the first 4 patients completed study activities, the investigator determined that this protocol is not the best way to test the study hypothesis due to uninterpretable data. Study was then terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT05128682/Prot_SAP_001.pdf